CLINICAL TRIAL: NCT02544763
Title: A Double-blind, Randomized, Placebo-controlled Study to Investigate the Efficacy and Safety of Cannabidiol (GWP42003-P, CBD) as Add-on Therapy in Patients With Tuberous Sclerosis Complex Who Experience Inadequately-controlled Seizures
Brief Title: A Randomized Controlled Trial of Cannabidiol (GWP42003-P, CBD) for Seizures in Tuberous Sclerosis Complex (GWPCARE6)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWEP1521 Blinded Phase; 2015-002154-12 (EudraCT Number)
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Tuberous Sclerosis Complex; Seizures
MeSH Terms: conditions — Tuberous Sclerosis; Seizures | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 25 mg/kg/day GWP42003-P (Experimental): 100 mg/mL GWP42003-P oral solution taken twice daily (morning and evening).
  Interventions: Drug: GWP42003-P
- 50 mg/kg/day GWP42003-P (Experimental): 100 mg/mL GWP42003-P oral solution taken twice daily (morning and evening).
  Interventions: Drug: GWP42003-P
- Placebo (Placebo Comparator): Placebo oral solution matching 100 mg/mL GWP42003-P.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GWP42003-P — Yellow oily solution containing cannabidiol dissolved in the excipients sesame oil and anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring.
  Other Names: Cannabidiol; CBD
  Arms: 25 mg/kg/day GWP42003-P; 50 mg/kg/day GWP42003-P
Drug: Placebo — Yellow oily solution containing the excipients sesame oil and anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring.
  Arms: Placebo

SUMMARY:
This trial consists of 2 parts: a double-blinded phase and an open-label extension phase. The blinded phase only will be described in this record. Participants will receive 1 of 2 doses of GWP42003-P or matching placebo. The primary clinical hypothesis is that there will be a difference between GWP42003-P and placebo in their effect on seizure frequency.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has a well-documented clinical history of epilepsy.
* Participant has a clinical diagnosis of Tuberous Sclerosis Complex (TSC) according to the criteria agreed by the 2012 International TSC Consensus Conference.
* All medications or interventions for epilepsy (including ketogenic diet and any neurostimulation devices for epilepsy) must have been stable for 1 month prior to screening and the participant is willing to maintain a stable regimen throughout the trial.

Key Exclusion Criteria:

* Participant has a history of pseudo-seizures.
* Participant has clinically significant unstable medical conditions other than epilepsy.
* Participant has an illness in the 4 weeks prior to screening or randomization, other than epilepsy, which in the opinion of the investigator could affect seizure frequency.
* Participant has undergone general anesthetic in the 4 weeks prior to screening or randomization.
* Participant has undergone surgery for epilepsy in the 6 months prior to screening.
* Participant is being considered for epilepsy surgery or any procedure involving general anesthesia.
* Participant has been taking felbamate for less than 1 year prior to screening.
* Participant is taking an oral mTOR inhibitor.
* Participant has any known or suspected hypersensitivity to cannabinoids or any of the excipients of the Investigational Medicinal Product (IMP), such as sesame oil.
* Participant has any history of suicidal behavior or any suicidal ideation of type 4 or 5 on the C-SSRS in the last month or at screening.
* Participant is currently using or has in the past used recreational or medicinal cannabis, or cannabinoid-based medications, within the 3 months prior to screening and is unwilling to abstain for the duration for the study.
* Participant has tumor growth which, in the opinion of the Investigator, could affect the primary endpoint.
* Participant has significantly impaired hepatic function at the screening or randomization visit
* Participant has received an IMP within the 12 weeks prior to the screening visit.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2016-04-06 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-02-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (23):
  - UAB Epilepsy Center, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UCLA-Pediatric Neurology, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University of Colorado Denver, Aurora, Colorado
  - Pediatric Neurology, Miami, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Mid Atlantic Epilepsy & Sleep Centre, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Minnesota Epilepsy Group, P.A, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Comprehensive Epilepsy Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - WellSpan Paediatric Neurology, Manchester, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Texas Scottish Rite Hospital for Children, Dallas, Texas
  - Cook Children's Health Care System, Fort Worth, Texas
  - Paediatric Neurology, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Australia (4):
  - Austin Health, Heidelberg
  - Royal Brisbane and Women's Hospital, Herston
  - The Royal Melbourne Hospital, Parkville
  - Sydney Children's Hospital, Randwick
- Netherlands (2):
  - Erasmus MC/Sophia Children's Hospital, Rotterdam
  - UMC Utrecht/ Wilhelmina, Kinderziekenhuis, Utrecht
- Poland (6):
  - Vitamed Gałaj I Cichomski Spółka Jawna, Bydgoszcz
  - Centrum Medyczne Plejady, Krakow
  - Wojewódzki Szpital Specjalistyczny im S. K. Wyszyńskiego SPZOZ, Lublin
  - Instytut "Pomnik - Centrum Zdrowia Dziecka", Warsaw
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego w Warszawie, Warsaw
  - Centrum Neuropsychiatrii "Neuromed", Wroclaw
- Spain (5):
  - Centro Médico Teknon, Barcelona
  - Clinical Research Unit, Barcelona
  - Unitat d'Epilèpsia, Barcelona
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Clinica Universidad de Navarra, Pamplona
- United Kingdom (4):
  - Cardiff and Vale University Local Health Board, Cardiff
  - Children and Young Adults' Research Unit, Cardiff
  - NIHR Clinical Research Facility, London
  - St George's University Hospitals NHS Foundation Trust, London

REFERENCES:
- [Derived] Burke C, Crossan C, Tyas E, Hemstock M, Lee D, Bowditch S. A Cost-Utility Analysis of Add-On Cannabidiol Versus Usual Care Alone for the Treatment of Seizures Associated with Tuberous Sclerosis Complex in England and Wales. Pharmacoecon Open. 2024 Jul;8(4):611-626. doi: 10.1007/s41669-024-00474-x. Epub 2024 Mar 5. PMID 38441854
- [Derived] Wu JY, Cock HR, Devinsky O, Joshi C, Miller I, Roberts CM, Sanchez-Carpintero R, Checketts D, Sahebkar F. Time to onset of cannabidiol treatment effect and resolution of adverse events in tuberous sclerosis complex: Post hoc analysis of randomized controlled phase 3 trial GWPCARE6. Epilepsia. 2022 May;63(5):1189-1199. doi: 10.1111/epi.17199. Epub 2022 Mar 4. PMID 35175622
- [Derived] Thiele EA, Bebin EM, Filloux F, Kwan P, Loftus R, Sahebkar F, Sparagana S, Wheless J. Long-term cannabidiol treatment for seizures in patients with tuberous sclerosis complex: An open-label extension trial. Epilepsia. 2022 Feb;63(2):426-439. doi: 10.1111/epi.17150. Epub 2021 Dec 27. PMID 34957550
- [Derived] Thiele EA, Bebin EM, Bhathal H, Jansen FE, Kotulska K, Lawson JA, O'Callaghan FJ, Wong M, Sahebkar F, Checketts D, Knappertz V; GWPCARE6 Study Group. Add-on Cannabidiol Treatment for Drug-Resistant Seizures in Tuberous Sclerosis Complex: A Placebo-Controlled Randomized Clinical Trial. JAMA Neurol. 2021 Mar 1;78(3):285-292. doi: 10.1001/jamaneurol.2020.4607. PMID 33346789

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 255 participants were screened; 31 of whom were screen failures. A total of 224 participants were randomized to double-blind treatment.
Groups:
- GWP42003-P 25 mg/kg/Day: Participants were randomized to receive GWP42003-P 25 milligrams per kilogram per day (mg/kg/day) (via oral twice daily [morning and evening] administration). Participants completed a 4-week dose escalation period, titrating up to their assigned dose, before continuing on a stable dose of blinded GWP42003-P for 12 weeks.
- GWP42003-P 50 mg/kg/Day: Participants were randomized to receive GWP42003-P 50 mg/kg/day (via oral twice daily [morning and evening] administration). Participants completed a 4-week dose escalation period, titrating up to their assigned dose, before continuing on a stable dose of blinded GWP42003-P for 12 weeks.
- Placebo: Participants were randomized to receive placebo matched to GWP42003-P (via oral twice daily [morning and evening] administration) for 16 weeks.
Period: Overall Study
Arm/Group | GWP42003-P 25 mg/kg/Day | GWP42003-P 50 mg/kg/Day | Placebo
Started | 75 | 73 | 76
Completed | 65 | 61 | 75
Not Completed | 10 | 12 | 1
Not completed — Adverse Event | 8 | 8 | 0
Not completed — Withdrawn by parent/guardian | 1 | 1 | 1
Not completed — Met withdrawal criteria | 0 | 2 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Difficulties taking IMP | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for members of the Safety Analysis Set, comprised of participants randomized to treatment who received at least 1 dose of investigational medicinal product (IMP).
Groups:
- Total: Total of all reporting groups
Arm/Group | GWP42003-P 25 mg/kg/Day | GWP42003-P 50 mg/kg/Day | Placebo | Total
Number analyzed (Participants) | 75 | 73 | 76 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Two participants were excluded from the summary of demographic data because their heights at screening were measured in inches but were recorded in centimeters.
  years
    number analyzed (Participants) | 75 | 72 | 75 | 222
    (all) | 14.112 (10.8131) | 12.915 (8.5324) | 13.918 (10.6302) | 13.659 (10.0324)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two participants were excluded from the summary of demographic data because their heights at screening were measured in inches but were recorded in centimeters.
  Participants
    number analyzed (Participants) | 75 | 72 | 75 | 222
    Female | 32 | 30 | 31 | 93
    Male | 43 | 42 | 44 | 129
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Two participants were excluded from the summary of demographic data because their heights at screening were measured in inches but were recorded in centimeters.
  Participants
    number analyzed (Participants) | 75 | 72 | 75 | 222
    White/Caucasian | 68 | 65 | 66 | 199
    Black/African American | 2 | 3 | 0 | 5
    American Indian/Alaska Native | 1 | 0 | 0 | 1
    Asian | 1 | 0 | 3 | 4
    Biracial Causasian-African American | 1 | 0 | 0 | 1
    Latin | 1 | 0 | 0 | 1
    Arabic | 1 | 0 | 0 | 1
    Caucasian/Asian | 0 | 1 | 0 | 1
    Hispanic/Latino | 0 | 2 | 0 | 2
    Hispanic | 0 | 1 | 3 | 4
    Hispanic And Caucasian | 0 | 0 | 1 | 1
    Anglo Indian | 0 | 0 | 1 | 1
    Black, White, American Indian | 0 | 0 | 1 | 1
Number of Tuberous Sclerosis Complex (TSC)-Associated Seizures [Mean (Standard Deviation); unit: seizures] — TSC-associated seizures included: focal motor seizures without impairment of consciousness or awareness (Type 1 focal motor); focal seizures with impairment of consciousness or awareness (Type 2 focal); focal seizures evolving to bilateral generalized convulsive seizures (Type 3 focal); and tonic-clonic, tonic, clonic, or atonic seizures that are countable. Population: Intent-to-Treat (ITT) Analysis Set: all participants who were randomized and dosed with IMP in the trial and had post-Baseline efficacy data. Participant data were analyzed according to the treatment group to which they were randomized.
  seizures | 77.95 (83.390) | 92.95 (89.782) | 89.22 (101.778) | 86.66 (91.841)
Number of Total Seizures [Mean (Standard Deviation); unit: seizures] — Total seizures included all seizure types combined. The Baseline Period included all data prior to Day 1. Population: ITT Analysis Set
  seizures | 80.87 (84.676) | 108.06 (115.699) | 118.32 (211.868) | 102.44 (148.495)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in the Number of Tuberous Sclerosis Complex (TSC)-Associated Seizures During the Treatment Period (Maintenance and Titration)
Description: TSC-associated seizures included: focal motor seizures without impairment of consciousness or awareness (Type 1 focal motor); focal seizures with impairment of consciousness or awareness (Type 2 focal); focal seizures evolving to bilateral generalized convulsive seizures (Type 3 focal); and tonic-clonic, tonic, clonic, or atonic seizures that are countable. Percent change from Baseline was calculated as the (post-Baseline value minus the Baseline value) divided by the Baseline value x 100.
Time Frame: Baseline; up to Week 16
Population: Intent-to-Treat (ITT) Analysis Set: all participants who were randomized and dosed with investigational medicinal product (IMP) in the trial and had post-Baseline efficacy data. Participant data were analyzed according to the treatment group to which they were randomized.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | GWP42003-P 25 mg/kg/Day | GWP42003-P 50 mg/kg/Day | Placebo
Number analyzed (Participants) | 75 | 73 | 76
percent change | -43.36 [-67.8 to -13.6] | -36.55 [-67.0 to -5.5] | -20.08 [-47.1 to 3.1]
Statistical Analysis 1: Comparison: GWP42003-P 25 mg/kg/Day; Test type: Superiority; Percentage reduction = 48.6, 95% CI 2-sided [40.4 to 55.8]
Statistical Analysis 2: Comparison: GWP42003-P 50 mg/kg/Day; Test type: Superiority; Percentage reduction = 47.5, 95% CI 2-sided [39.0 to 54.8]
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority; Percentage reduction = 26.5, 95% CI 2-sided [14.9 to 36.5]
Statistical Analysis 4: Comparison: GWP42003-P 25 mg/kg/Day vs Placebo; Test type: Superiority; p = 0.0009, Mixed Models Analysis; Treatment ratio = 0.699, 95% CI 2-sided [0.567 to 0.861]
Statistical Analysis 5: Comparison: GWP42003-P 50 mg/kg/Day vs Placebo; Test type: Superiority; p = 0.0018, Mixed Models Analysis; Treatment ratio = 0.715, 95% CI 2-sided [0.580 to 0.881]

2. Secondary Outcome: Number of Participants Considered Treatment Responders During the Treatment Period (Maintenance and Titration)
Description: Treatment responders are defined as those participants with a ≥ 50% reduction in TSC-associated seizure frequency. TSC-associated seizures included: focal motor seizures without impairment of consciousness or awareness (Type 1 focal motor); focal seizures with impairment of consciousness or awareness (Type 2 focal); focal seizures evolving to bilateral generalized convulsive seizures (Type 3 focal); and tonic-clonic, tonic, clonic, or atonic seizures that are countable. Participants who withdrew from the trial during the treatment period are considered non-responders.
Time Frame: Baseline; up to Week 16
Population: ITT Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P 25 mg/kg/Day | GWP42003-P 50 mg/kg/Day | Placebo
Number analyzed (Participants) | 75 | 73 | 76
Participants
  Responders | 27 | 29 | 17
  Non-responders | 48 | 44 | 59
Statistical Analysis 1: Comparison: GWP42003-P 25 mg/kg/Day vs Placebo; Test type: Superiority; p = 0.0692, Cochran-Mantel-Haenszel; The p-value was calculated from a Cochran-Mantel-Haenszel test stratified by age group (1-6, 7-11, 12-17 and 18-65 years); Odds Ratio (OR) = 1.95, 95% CI 2-sided [0.95 to 4.00]
Statistical Analysis 2: Comparison: GWP42003-P 50 mg/kg/Day vs Placebo; Test type: Superiority; p = 0.0245, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.29, 95% CI 2-sided [1.12 to 4.67]

3. Secondary Outcome: Change From Baseline in the Caregiver Global Impression of Change (CGIC) or Participant Global Impression of Change (PGIC) Score at the Participant's Last Visit
Description: The combined caregiver and participant summary uses either the caregiver or participant version if only one version was completed, or the caregiver version if both caregiver and participant versions were completed. The CGIC comprised the following question, to be rated on a 7-point scale (1, Very Much Improved; 2, Much Improved; 3, Slightly Improved; 4, No Change; 5, Slightly Worse; 6, Much Worse; 7, Very Much Worse): "Since your child started treatment, please assess the status of your child's overall condition (comparing their condition now to their condition before treatment)." The SGIC comprised the following question, to be rated on a 7-point scale (1, Very Much Improved; 2, Much Improved; 3, Slightly Improved; 4, No Change; 5, Slightly Worse; 6, Much Worse; 7, Very Much Worse): "Since you started treatment, please assess the status of your overall condition (comparing your condition now to your condition before treatment)."
Time Frame: Baseline; up to Week 16
Population: ITT Analysis Set. Only participants with available data were analyzed. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003-P 25 mg/kg/Day | GWP42003-P 50 mg/kg/Day | Placebo
Number analyzed (Participants) | 75 | 73 | 76
units on a scale
  Caregiver: number analyzed (Participants) | 66 | 66 | 72
  Caregiver | 3.0 (1.34) | 3.1 (1.40) | 3.5 (0.93)
  Combined Caregiver and Participant: number analyzed (Participants) | 70 | 69 | 76
  Combined Caregiver and Participant | 3.0 (1.35) | 3.2 (1.45) | 3.5 (0.96)
  Participant: number analyzed (Participants) | 6 | 4 | 4
  Participant | 3.3 (1.51) | 4.5 (1.73) | 2.8 (1.26)
Statistical Analysis 1: Comparison: GWP42003-P 25 mg/kg/Day vs Placebo; Test type: Superiority; p = 0.0074, nominal; The global impression of change was analyzed using an ordinal logistic regression model with treatment group as a fixed factor; Odds Ratio (OR) = 2.25, 95% CI 2-sided [1.24 to 4.07]
Statistical Analysis 2: Comparison: GWP42003-P 50 mg/kg/Day vs Placebo; Test type: Superiority; p = 0.0580, nominal; The global impression of change is analyzed using an ordinal logistic regression model with treatment group as a fixed factor; Odds Ratio (OR) = 1.77, 95% CI 2-sided [0.98 to 3.20]

4. Secondary Outcome: Percent Change From Baseline in Total Seizures During the Treatment Period (Maintenance and Titration)
Description: Total seizures included all seizure types combined. Percent change from Baseline was calculated as the (post-Baseline value minus the Baseline value) divided by the Baseline value x 100.
Time Frame: Baseline; up to Week 16
Population: ITT Analysis Set
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | GWP42003-P 25 mg/kg/Day | GWP42003-P 50 mg/kg/Day | Placebo
Number analyzed (Participants) | 75 | 73 | 76
percent change | -34.71 (46.150) | -35.14 (42.530) | -19.63 (35.137)
Statistical Analysis 1: Comparison: GWP42003-P 25 mg/kg/Day; Test type: Superiority — Model includes the total number of seizures as a response variable and age group, time (Baseline and treatment period), treatment and treatment by time interaction as fixed effects and participant as a random effect. The log transformed number of days seizures were reported by period is included as an offset; Percentage reduction = 0.519, 95% CI 2-sided [0.447 to 0.602]
Statistical Analysis 2: Comparison: GWP42003-P 50 mg/kg/Day; Test type: Superiority; Percentage reduction = 0.524, 95% CI 2-sided [0.452 to 0.607]
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority; Percentage reduction = 0.731, 95% CI 2-sided [0.632 to 0.846]
Statistical Analysis 4: Comparison: GWP42003-P 25 mg/kg/Day vs Placebo; Test type: Superiority; p = 0.0013, Mixed Models Analysis; Treatment ratio = 0.709, 95% CI 2-sided [0.576 to 0.873]
Statistical Analysis 5: Comparison: GWP42003-P 50 mg/kg/Day vs Placebo; Test type: Superiority; p = 0.0018, Mixed Models Analysis; Treatment ratio = 0.716, 95% CI 2-sided [0.582 to 0.882]

5. Secondary Outcome: Number of Participants With Any Severe Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as an AE with a start date on or after the first dose of IMP during the Blinded Phase up to and including the date of first dose of the Open-label Extension (OLE) Phase (OLE Day 1).
Time Frame: up to approximately Week 22
Population: Safety Analysis Set: all participants randomized to treatment who received at least 1 dose of IMP
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P 25 mg/kg/Day | GWP42003-P 50 mg/kg/Day | Placebo
Number analyzed (Participants) | 75 | 73 | 76
Participants | 7 | 9 | 1

ADVERSE EVENTS:
Time Frame: up to approximately Week 22
Description: Baseline data are reported for members of the Safety Analysis Set, comprised of participants randomized to treatment who received at least 1 dose of investigational medicinal product (IMP). Treatment-emergent adverse events are defined as adverse events with a start date on or after the first dose of IMP during the Blinded Phase up to and including the date of the first dose of the Open-label Extension (OLE) Phase (OLE Day 1).
Arm/Group | GWP42003-P 25 mg/kg/Day | GWP42003-P 50 mg/kg/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/73 | 0/76
Serious Adverse Events (participants affected / at risk) | 16/75 | 10/73 | 2/76
Other Adverse Events (participants affected / at risk) | 66/75 | 71/73 | 68/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GWP42003-P 25 mg/kg/Day (N=75) | GWP42003-P 50 mg/kg/Day (N=73) | Placebo (N=76)
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Type IV hypersensitivity reaction (Immune system disorders) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 0
Transaminases increased (Investigations) | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 2 | 0 | 1
Seizure (Nervous system disorders) | 1 | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P 25 mg/kg/Day (N=75) | GWP42003-P 50 mg/kg/Day (N=73) | Placebo (N=76)
Anaemia (Blood and lymphatic system disorders) | 5 | 3 | 1
Ear pain (Ear and labyrinth disorders) | 2 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 1
Constipation (Gastrointestinal disorders) | 8 | 5 | 6
Diarrhoea (Gastrointestinal disorders) | 23 | 40 | 19
Frequent bowel movements (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 6 | 2 | 2
Retching (Gastrointestinal disorders) | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 12 | 13 | 7
Fatigue (General disorders) | 3 | 4 | 1
Gait disturbance (General disorders) | 4 | 3 | 2
Pyrexia (General disorders) | 14 | 12 | 6
Bronchitis (Infections and infestations) | 2 | 1 | 1
Ear infection (Infections and infestations) | 2 | 4 | 0
Gastroenteritis (Infections and infestations) | 3 | 2 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 3 | 3
Nasopharyngitis (Infections and infestations) | 11 | 11 | 12
Otitis media (Infections and infestations) | 2 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 2 | 2
Pharyngitis streptococcal (Infections and infestations) | 0 | 2 | 1
Pneumonia (Infections and infestations) | 2 | 2 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 2
Tonsillitis (Infections and infestations) | 2 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 7 | 10
Urinary tract infection (Infections and infestations) | 4 | 1 | 0
Viral infection (Infections and infestations) | 3 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 4 | 5
Laceration (Injury, poisoning and procedural complications) | 0 | 2 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 2 | 1
Alanine aminotransferase increased (Investigations) | 7 | 14 | 0
Anticonvulsant drug level increased (Investigations) | 1 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 12 | 0
Eosinophil count increased (Investigations) | 4 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 12 | 10 | 0
Hepatic enzyme increased (Investigations) | 0 | 3 | 0
International normalised ratio increased (Investigations) | 0 | 2 | 0
Platelet count decreased (Investigations) | 3 | 2 | 0
Prothrombin time prolonged (Investigations) | 0 | 2 | 0
Weight decreased (Investigations) | 5 | 6 | 0
Decreased appetite (Metabolism and nutrition disorders) | 15 | 17 | 9
Diet refusal (Metabolism and nutrition disorders) | 0 | 2 | 0
Increased appetite (Metabolism and nutrition disorders) | 3 | 3 | 5
Ataxia (Nervous system disorders) | 3 | 2 | 2
Dizziness (Nervous system disorders) | 2 | 0 | 3
Drooling (Nervous system disorders) | 1 | 2 | 2
Headache (Nervous system disorders) | 4 | 2 | 4
Hypersomnia (Nervous system disorders) | 0 | 2 | 0
Lethargy (Nervous system disorders) | 4 | 3 | 5
Seizure (Nervous system disorders) | 4 | 7 | 5
Somnolence (Nervous system disorders) | 10 | 19 | 7
Abnormal behaviour (Psychiatric disorders) | 1 | 2 | 1
Aggression (Psychiatric disorders) | 2 | 2 | 3
Agitation (Psychiatric disorders) | 1 | 2 | 3
Anxiety (Psychiatric disorders) | 2 | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 2 | 5
Irritability (Psychiatric disorders) | 4 | 5 | 4
Panic attack (Psychiatric disorders) | 2 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 7 | 2
Hypertension (Vascular disorders) | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT02544763/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT02544763/SAP_001.pdf